CLINICAL TRIAL: NCT03663491
Title: Necessity of Transnasal Gastroscopy in Routine Diagnostics - a Patient Centered Requirement Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Nasal Gastroscopy
Record Dates: First submitted 2018-06-21; First posted 2018-09-10 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2018-05

CONDITIONS: Patient Safety
Keywords: Gastroscopy; Transnasal Endoscopy; Sedation
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Unsedated Nasal Gastroscopy (Experimental): Transnasal Endoscopy. No sedation used. Use of local anesthesia.
  Interventions: Procedure: Nasal Gastroscopy; Procedure: Oral Gastroscopy with transnasal endoscope, sedated
- Oral Gastroscopy, unsedated (Active Comparator): Transoral Endoscopy. No sedation used. Use of local anesthesia.
  Interventions: Procedure: Oral Gastroscopy, unsedated
- Oral Gastroscopy, sedated (Active Comparator): Transoral Endoscopy. Intravenous sedation used.
  Interventions: Procedure: Oral Gastroscopy, sedated

INTERVENTIONS:
Procedure: Nasal Gastroscopy — Use of transnasal endoscopes for routine gastroscopy in adults.
  Arms: Unsedated Nasal Gastroscopy
Procedure: Oral Gastroscopy, unsedated — Use of transoral endoscopes for routine gastroscopy in adults. Use of local anesthesia.
  Arms: Oral Gastroscopy, unsedated
Procedure: Oral Gastroscopy, sedated — Use of transoral endoscopes for routine gastroscopy in adults. Use of intravenous sedation.
  Arms: Oral Gastroscopy, sedated
Procedure: Oral Gastroscopy with transnasal endoscope, sedated — Use of transnasal endoscopes for routine gastroscopy in adults, following a failed attempt to perform transnasal gastroscopy
  Arms: Unsedated Nasal Gastroscopy

SUMMARY:
Evaluation of patients safety and comfort in nasal endoscopy.

DETAILED DESCRIPTION:
Introduction: Numerous indications require regular outpatient upper gastrointestinal endoscopy (EGD). In most cases, peroral gastroscopy is performed. The aim of this study was to evaluate the necessity and outpatients' demand for transnasal gastroscopy (nEGD).

Methods: A questionnaire was used to assess patients' choice of method, previous experience, psychological and sociodemographic data. Furthermore, the patients' satisfaction with and potentially perceived discomfort during the examination as well as their preference for a method with regard to future examinations was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Adequate knowledge of oral and written german

Exclusion Criteria:

* Inpatient Treatment
* For medical reasons (narrow nasal cavity, band ligation of esophageal varices, Placement of a percutaneous endoscopic gastrostomy, planned colonoscopy under sedation the same day, abnormal coagulation, emergency procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Patients satisfaction (pain, discomfort, experience) | During Endoscopy procedure
  Satisfaction with the procedure:
  * not at all
  * hardly
  * moderately
  * quite
  * extraordinarily
  (extraordinarily = the best possible outcome, not at all = the worst possible outcome)

SECONDARY OUTCOMES:
Pain during the procedure | During Endoscopy procedure
  Nose pain Numeric Rating Scale 1-10 (1 = no pain, 10 = worst imaginable pain)
  Throat pain Numeric Rating Scale 1-10 (1 = no pain, 10 = worst imaginable pain)
  Gag Reflex:
  Yes or No
  Abdominal pain:
  Numeric Rating Scale 1-10 (1 = no pain, 10 = worst imaginable pain)
Previous experience with endoscopy | Before Endoscopy procedure
  Experience:
  Have you had a gastroscopy:
  Yes or No
  If Yes, how was your gastroscopy:
  * pleasant
  * slightly unpleasant
  * very unpleasant

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Hoffmeister, Prof Dr, Study Chair — University of Leipzig
Locations (1):
- University of Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Yes
All data will be available to other researchers on request. (Mail to juergen.feisthammel@medizin.uni-leipzig.de)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be available to other researchers on request. (Mail to juergen.feisthammel@medizin.uni-leipzig.de)
Access Criteria: All data will be available to other researchers on request. (Mail to juergen.feisthammel@medizin.uni-leipzig.de)

REFERENCES:
- [Derived] Schuldt AL, Kirsten H, Tuennemann J, Heindl M, van Bommel F, Feisthammel J, Hollenbach M, Hoffmeister A. Necessity of transnasal gastroscopy in routine diagnostics: a patient-centred requirement analysis. BMJ Open Gastroenterol. 2019 Apr 14;6(1):e000264. doi: 10.1136/bmjgast-2018-000264. eCollection 2019. PMID 31139423